CLINICAL TRIAL: NCT03176784
Title: UW Quitting Using Intensive Treatment Study
Brief Title: UW Quitting Using Intensive Treatment Study (QUITS)
Acronym: QUITS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Washington University School of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0404; R01HL109031 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 6/11/2020 (Other: UW Madison)
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Tobacco Dependence
Keywords: Varenicline; Nicotine Patch; Quit Smoking; Tobacco; Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Intervention Model Description: Double Blinded Placebo Controlled Factorial
Who Masked: Participant, Care Provider
Masking Description: Active and placebo medications are identical in appearance. Medication labeling and the dispensing protocol are designed to prevent participants and care providers from knowing if the medication is active or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Varenicline + Patch Standard Duration (Experimental): Standard Condition Varenicline: 0.5 mg pill once daily (QD) on Days -7 to -5; 0.5 mg pill twice daily (BID) Days -4 to -1; 1 mg pill BID Days 1 to Week 11; Placebo Pill weeks 12-23 BID
  Standard Condition Nicotine Patches:
  Patches (Nicotine): 14 mg Patches for 2 weeks prequit and then 10 weeks post-quit, then 7 mg patches for Weeks 11 and 12; Placebo patches weeks 13-24
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Other: Placebo Patch; Other: Placebo Pill
- Varenicline Only Standard Duration (Experimental): Standard Condition Varenicline: 0.5 mg pill QD on Days -7 to -5; 0.5 mg pill BID Days -4 to -1; 1 mg pill BID Days 1 to Week 11; Placebo Pill weeks 12-23 BID
  Standard Condition Placebo Patches:
  Placebo patches for 2 weeks prequit and for weeks 1-24 post-quit
  Interventions: Drug: Varenicline; Other: Placebo Patch; Other: Placebo Pill
- Varenicline + Patch Extended Duration (Experimental): Extended Condition Varenicline: 0.5 mg pill QD on Days -7 to -5, 0.5 mg pill BID Days -4 to -1, and 1 mg pill BID Days 1 to Week 22
  Extended Condition Nicotine Patches:
  14 mg Patches for 2 weeks prequit and then weeks 1-22 post-quit, then 7 mg patches for Weeks 23 and 24 post-quit.
  Interventions: Drug: Varenicline; Drug: Nicotine patch
- Varenicline Only Extended Duration (Experimental): Extended Condition Varenicline: 0.5 mg pill QD on Days -7 to -5, 0.5 mg pill BID Days -4 to -1, and 1 mg pill BID Days 1 to Week 22
  Extended Condition Placebo Patches:
  Placebo patches for 2 weeks prequit and for weeks 1-24 post-quit
  Interventions: Drug: Varenicline; Other: Placebo Patch

INTERVENTIONS:
Drug: Varenicline — 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Other Names: Chantix
Drug: Nicotine patch — 14 mg and 7 mg nicotine patches used. See arms for specific durations.
  Other Names: Nicoderm CQ
  Arms: Varenicline + Patch Extended Duration; Varenicline + Patch Standard Duration
Other: Placebo Patch — Placebo patches matched in appearance to the Active 14 mg and 7 mg nicotine patches used in the Nicotine patch intervention. See arms for specific durations.
  Arms: Varenicline + Patch Standard Duration; Varenicline Only Extended Duration; Varenicline Only Standard Duration
Other: Placebo Pill — Placebo pills matched in appearance to the Active Varenicline pills in the Varenicline intervention. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Arms: Varenicline + Patch Standard Duration; Varenicline Only Standard Duration

SUMMARY:
This research will determine whether two highly promising modifications to varenicline treatment (i.e. use of a nicotine patch adjuvant and extended 24-week duration) produce superior smoking outcomes when they are either used together or alone. Despite their promise, the proposed modifications have never been experimentally evaluated relative to standard varenicline pharmacotherapy. Thus, this innovative research will produce novel evidence regarding how best to help smokers quit, and thereby address the leading cause of preventable mortality and morbidity related to cardiovascular and pulmonary diseases.

DETAILED DESCRIPTION:
Building on our recent NHLBI-funded publication in JAMA (see references below) that described the modest effectiveness of varenicline pharmacotherapy, this study will use a 2 X 2 factorial design to evaluate two different medication use strategies on their ability to markedly enhance varenicline effectiveness in a large cohort of current smokers. Smokers (N=1000) will be randomly assigned to one of two levels for each of two factors: 1) an Adjuvant factor (varenicline + placebo patch versus varenicline + nicotine patch), and 2) a Duration factor (12 versus 24 weeks of active medication). Thus, this factorial design yields a "standard" varenicline treatment (12 weeks of active varenicline and 12 weeks of placebo varenicline + 24 weeks of placebo patch), and 3 enhanced treatments: 1) 12 weeks of active varenicline and 12 weeks of placebo varenicline + 24 weeks of active patch, 2) 24-weeks of active varenicline + 24 weeks of placebo patch, and 3) 24 weeks of active varenicline + 24 weeks of active patch.

Both treatment modifications, longer duration therapy and use of a nicotine replacement therapy (NRT) adjuvant, have produced some quite promising effects. However, in both cases these modifications have been little researched, their effects are not consistently positive, and they have not been implemented in a potentially optimal manner. We will implement each modification in an innovative manner designed to enhance its effectiveness. In addition, all participants will be given counseling that supports adherent medication use and that is readily translatable to healthcare settings. The scientific rigor of this work will be enhanced by the use of placebo medication, a large sample, and a factorial design. The latter will allow us to test both the main and interaction effects of the experimental factors. We will also be able to compare each enhanced treatment with standard 12-week varenicline-only therapy to determine whether any of these medication use strategies significantly enhances treatment effectiveness.

ELIGIBILITY:
Inclusion criteria:

Participants must: plan to stay in the area for the next 12 months, ability to read and write in English, smoke on average ≥5 cigarettes per day over the last 6 months, be ≥18 years old, desire to quit smoking but not be engaged currently in cessation treatment, report no use of pipe tobacco, cigars, snuff, e-cigarettes or chew in the last 30 days, have reliable phone access, willing and able to use both nicotine patch and varenicline, access to transportation to come to our clinic and, if female, not be pregnant and be using an acceptable birth control method/ method to prevent pregnancy. Smoking will be biochemically confirmed via a carbon monoxide (CO) breath test at the orientation session visit. Potential participants must have a CO test result of ≥5ppm for eligibility to participate.

Exclusion criteria:

Current treatment for schizophrenia or a psychotic disorder; suicidal ideation in the past 12 months; history of suicidal attempts within the last 10 years; on dialysis or being told you have severe kidney disease; hospitalization for a stroke, heart attack, congestive heart failure or uncontrolled diabetes mellitus within the past year; history of seizure within the last year; currently taking Wellbutrin, Zyban, or Buproprion (Contrave is a weight-loss drug that has Wellbutrin in it) for reasons other than to quit smoking or taking to help quit smoking and not willing to stop for duration of the study; currently using any form of nicotine replacement (e.g., nicotine patch, nicotine gum, nicotine lozenge) or using Chantix or varenicline and not willing to stop for duration of the study; had a reaction to the nicotine patch that prevented them from continuing to use it; or currently participating in another smoking cessation study.

Pregnancy:

Even though we screen out participants who are pregnant, plan to become pregnant, nursing, or are unwilling to take steps to avoid pregnancy, there is a chance that a participant eligible at consent could become pregnant later. She would then be considered part of a vulnerable group. Given the longitudinal nature of the research, a participant who becomes pregnant after enrolling will be given the choice of whether to 1) continue in the study (for counseling and other assessments) and agree to immediately stop taking study meds for the remaining duration of the study and return any unused medications, OR 2) withdraw. No further medications will be given to this study participant while in the study.

Incarcerated Individuals:

Incarcerated individuals will not be enrolled in this study. However, given the longitudinal nature of the research, participants could be incarcerated for periods during their participation. If study staff learn that a participant is incarcerated at a time point before or at their Week 8 phone call, the participant will be withdrawn from the study. If study staff learn that a participant is incarcerated subsequent to Week 8, the participant will not be withdrawn unless that incarceration will take them beyond the study period. In that case, staff will not contact the participant while incarcerated and will not provide any treatment (counseling or medication) nor conduct any assessments during the period of incarceration. Services and assessments will be re-initiated if the participant is released at a later study time point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1251 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Center For Tobacco Research and Intervention, Madison, Wisconsin
  - UW Center for Tobacco Research and Intervention, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data set will be posted by UW-CTRI in accord with NHLBI policies
Time Frame: 12 months after publication of the primary outcome paper.
Access Criteria: Prior written data request to the PI.

REFERENCES:
- [Background] Baker TB, Piper ME, Stein JH, Smith SS, Bolt DM, Fraser DL, Fiore MC. Effects of Nicotine Patch vs Varenicline vs Combination Nicotine Replacement Therapy on Smoking Cessation at 26 Weeks: A Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):371-9. doi: 10.1001/jama.2015.19284. PMID 26813210
- [Derived] Baker TB, Piper ME, Smith SS, Bolt DM, Stein JH, Fiore MC. Effects of Combined Varenicline With Nicotine Patch and of Extended Treatment Duration on Smoking Cessation: A Randomized Clinical Trial. JAMA. 2021 Oct 19;326(15):1485-1493. doi: 10.1001/jama.2021.15333. PMID 34665204
- See also: UW Center for Tobacco Research and Intervention website — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred via community outreach (e.g., social networking sites, radio, TV, newspaper). Interested respondents were called and screened for initial eligibility; those eligible attended a group orientation session that entailed: final eligibility assessment, written informed consent, baseline assessments, biochemical confirmation of smoking status, and randomization. Study visits were in Madison and Milwaukee, WI. First participant enrolled on 11/11/17; study completed on 7/9/20.
Groups:
- Varenicline + Patch Standard Duration: Standard Condition Varenicline: 0.5 mg pill once daily (QD) on Days -7 to -5; 0.5 mg pill twice daily (BID) Days -4 to -1; 1 mg pill BID Days 1 to Week 11; Placebo Pill weeks 12-23 BID
  Standard Condition Nicotine Patches:
  Patches (Nicotine): 14 mg Patches for 2 weeks prequit and then 10 weeks post-quit, then 7 mg patches for Weeks 11 and 12; Placebo patches weeks 13-24
  Varenicline: 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Nicotine patch: 14 mg and 7 mg nicotine patches used. See arms for specific durations.
  Placebo Patch: Placebo patches matched in appearance to the Active 14 mg and 7 mg nicotine patches used in the Nicotine patch intervention. See arms for specific durations.
  Placebo Pill: Placebo pills matched in appearance to the Active Varenicline pills in the Varenicline intervention. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
- Varenicline Only Standard Duration: Standard Condition Varenicline: 0.5 mg pill QD on Days -7 to -5; 0.5 mg pill BID Days -4 to -1; 1 mg pill BID Days 1 to Week 11; Placebo Pill weeks 12-23 BID
  Standard Condition Placebo Patches:
  Placebo patches for 2 weeks prequit and for weeks 1-24 post-quit
  Varenicline: 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Placebo Patch: Placebo patches matched in appearance to the Active 14 mg and 7 mg nicotine patches used in the Nicotine patch intervention. See arms for specific durations.
  Placebo Pill: Placebo pills matched in appearance to the Active Varenicline pills in the Varenicline intervention. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
- Varenicline + Patch Extended Duration: Extended Condition Varenicline: 0.5 mg pill QD on Days -7 to -5, 0.5 mg pill BID Days -4 to -1, and 1 mg pill BID Days 1 to Week 22
  Extended Condition Nicotine Patches:
  14 mg Patches for 2 weeks prequit and then weeks 1-22 post-quit, then 7 mg patches for Weeks 23 and 24 post-quit.
  Varenicline: 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Nicotine patch: 14 mg and 7 mg nicotine patches used. See arms for specific durations.
- Varenicline Only Extended Duration: Extended Condition Varenicline: 0.5 mg pill QD on Days -7 to -5, 0.5 mg pill BID Days -4 to -1, and 1 mg pill BID Days 1 to Week 22
  Extended Condition Placebo Patches:
  Placebo patches for 2 weeks prequit and for weeks 1-24 post-quit
  Varenicline: 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Placebo Patch: Placebo patches matched in appearance to the Active 14 mg and 7 mg nicotine patches used in the Nicotine patch intervention. See arms for specific durations.
Period: Overall Study
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
Started | 314 | 315 | 311 | 311
Completed | 209 | 202 | 198 | 241
Not Completed | 105 | 113 | 113 | 70
Not completed — Lost to Follow-up | 77 | 79 | 79 | 49
Not completed — Withdrawal by Subject | 28 | 34 | 34 | 21

BASELINE CHARACTERISTICS:
Groups:
- Varenicline + Patch Standard Duration: Standard Condition Varenicline: 0.5 mg pill QD on Days -7 to -5; 0.5 mg pill BID Days -4 to -1; 1 mg pill BID Days 1 to Week 11; Placebo Pill weeks 12-23 BID
  Standard Condition Nicotine Patches:
  Patches (Nicotine): 14 mg Patches for 2 weeks prequit and then 10 weeks post-quit, then 7 mg patches for Weeks 11 and 12; Placebo patches weeks 13-24
  Varenicline: 0.5mg and 1.0 mg pills used. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
  Nicotine patch: 14 mg and 7 mg nicotine patches used. See arms for specific durations.
  Placebo Patch: Placebo patches matched in appearance to the Active 14 mg and 7 mg nicotine patches used in the Nicotine patch intervention. See arms for specific durations.
  Placebo Pill: Placebo pills matched in appearance to the Active Varenicline pills in the Varenicline intervention. See arms for specific durations. (Active and placebo varenicline pills provided at no cost through an independent research agreement with Pfizer.)
- Total: Total of all reporting groups
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration | Total
Number analyzed (Participants) | 314 | 315 | 311 | 311 | 1251
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.4) | 48.6 (11.4) | 48.9 (12.3) | 49.9 (11.5) | 49.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 171 | 166 | 167 | 675
  Male | 143 | 144 | 145 | 144 | 576
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 12 | 5 | 41
  Not Hispanic or Latino | 285 | 297 | 285 | 297 | 1164
  Unknown or Not Reported | 15 | 8 | 14 | 9 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 4 | 2 | 14
  Asian | 2 | 2 | 3 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 2 | 3
  Black or African American | 71 | 70 | 68 | 78 | 287
  White | 221 | 219 | 213 | 214 | 867
  More than one race | 5 | 6 | 9 | 7 | 27
  Unknown or Not Reported | 12 | 12 | 14 | 7 | 45
Region of Enrollment [Number; unit: participants]
  United States | 314 | 315 | 311 | 311 | 1251

OUTCOME MEASURES:

1. Primary Outcome: 52-Week Point-Prevalence Abstinence
Description: Biochemically-confirmed self-reported total abstinence from any cigarette use (even a single puff) for the seven days preceding the target follow-up day, confirmed with an exhaled carbon monoxide reading of less than or equal to 5 ppm.
Time Frame: Assessed 52 weeks after quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
Number analyzed (Participants) | 314 | 315 | 311 | 311
Participants | 74 | 79 | 78 | 76
Statistical Analysis 1: Comparison: Varenicline + Patch Standard Duration vs Varenicline Only Standard Duration; Test type: Superiority; p = .66, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.6 to 1.3]
Statistical Analysis 2: Comparison: Varenicline Only Standard Duration vs Varenicline Only Extended Duration; Test type: Superiority; p = .85, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.4]
Statistical Analysis 3: Comparison: Varenicline Only Standard Duration vs Varenicline + Patch Extended Duration; Test type: Superiority; p = 1.00, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.4]

2. Secondary Outcome: 23-Week Point-Prevalence Abstinence
Description: Biochemically confirmed self-reported total abstinence from any cigarette use (even a single puff) for the seven days preceding the target follow-up day, confirmed with an exhaled carbon monoxide reading of less than or equal to 5 ppm.
Time Frame: Assessed 23 weeks after quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
Number analyzed (Participants) | 314 | 315 | 311 | 311
Participants | 74 | 66 | 82 | 70
Statistical Analysis 1: Comparison: Varenicline + Patch Standard Duration vs Varenicline Only Standard Duration; Test type: Superiority; p = .44, Regression, Logistic — Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.8 to 1.7]
Statistical Analysis 2: Comparison: Varenicline Only Standard Duration vs Varenicline Only Extended Duration; Test type: Superiority; p = .61, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.8 to 1.6]
Statistical Analysis 3: Comparison: Varenicline Only Standard Duration vs Varenicline + Patch Extended Duration; Test type: Superiority; p = .12, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.0]

3. Secondary Outcome: 52-Week Prolonged Abstinence
Description: Biochemically confirmed self-reported total abstinence from any cigarette use (even a single puff) from week 2 post-quit through week 52 post-quit, confirmed with an exhaled carbon monoxide reading of less than or equal to 5 ppm.
Time Frame: Assessed 52 weeks after quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
Number analyzed (Participants) | 314 | 315 | 311 | 311
Participants | 47 | 55 | 57 | 46
Statistical Analysis 1: Comparison: Varenicline + Patch Standard Duration vs Varenicline Only Standard Duration; Test type: Superiority; p = .43, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 2: Comparison: Varenicline Only Standard Duration vs Varenicline Only Extended Duration; Test type: Superiority; p = .37, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 3: Comparison: Varenicline Only Standard Duration vs Varenicline + Patch Extended Duration; Test type: Superiority; p = .81, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.6]

4. Secondary Outcome: 23-Week Prolonged Abstinence
Description: Biochemically confirmed self-reported total abstinence from any cigarette use (even a single puff) from week 2 post-quit through week 23 post-quit, confirmed with an exhaled carbon monoxide reading of less than or equal to 5 ppm.
Time Frame: Assessed 23 weeks after quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
Number analyzed (Participants) | 314 | 315 | 311 | 311
Participants | 66 | 72 | 73 | 65
Statistical Analysis 1: Comparison: Varenicline + Patch Standard Duration vs Varenicline Only Standard Duration; Test type: Superiority; p = .65, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.6 to 1.3]
Statistical Analysis 2: Comparison: Varenicline Only Standard Duration vs Varenicline Only Extended Duration; Test type: Superiority; p = .60, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.6 to 1.3]
Statistical Analysis 3: Comparison: Varenicline Only Standard Duration vs Varenicline + Patch Extended Duration; Test type: Superiority; p = .86, Regression, Logistic; Study site (Madison vs Milwaukee) was included as a covariate; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected and tabulated for the first 12 weeks of treatment.
Description: Some participants did not complete the adverse event assessments. The denominators used to calculate the percentage of participants reporting a given adverse event in each of the four conditions equal the number of participants responding to the adverse event assessment inquiry. Thus, the denominators do not equal the number of participants who started the study in each of the four conditions.
Arm/Group | Varenicline + Patch Standard Duration | Varenicline Only Standard Duration | Varenicline + Patch Extended Duration | Varenicline Only Extended Duration
All-Cause Mortality (participants affected / at risk) | 0/314 | 0/315 | 0/311 | 0/311
Serious Adverse Events (participants affected / at risk) | 0/314 | 1/315 | 0/311 | 1/311
Other Adverse Events (participants affected / at risk) | 194/305 | 164/300 | 159/295 | 160/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline + Patch Standard Duration (N=314) | Varenicline Only Standard Duration (N=315) | Varenicline + Patch Extended Duration (N=311) | Varenicline Only Extended Duration (N=311)
Anaphylaxis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline + Patch Standard Duration (N=305) | Varenicline Only Standard Duration (N=300) | Varenicline + Patch Extended Duration (N=295) | Varenicline Only Extended Duration (N=307)
Nausea (Gastrointestinal disorders) | 92 (92) | 72 (72) | 73 (73) | 95 (95)
Headache (Nervous system disorders) | 12 (12) | 20 (20) | 16 (16) | 17 (17)
Itching/Hives (Skin and subcutaneous tissue disorders) | 40 (40) | 9 (9) | 39 (39) | 14 (14)
Skin Rash (Skin and subcutaneous tissue disorders) | 53 (53) | 34 (34) | 51 (51) | 30 (30)
Insomnia (Psychiatric disorders) | 93 (93) | 88 (88) | 72 (72) | 83 (83)
Changes in Mood (Psychiatric disorders) | 50 (50) | 48 (48) | 53 (53) | 50 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03176784/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT03176784/ICF_001.pdf